CLINICAL TRIAL: NCT06220617
Title: Multi-omics Study for Early Detection of Colorectal Cancer Based on Liquid Biopsy Technology
Brief Title: Multi-omics Study for Early Detection of Colorectal Cancer (MOED-CRC)
Status: Recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Collaborators: New Horizon Health Technology Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Ding Ke-Feng, Chief physician, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: MOED-CRC
Record Dates: First submitted 2024-01-14; First posted 2024-01-24 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Cancer; Adenomatous Polyps; Adenoma; Advanced Adenoma
Keywords: Colorectal Cancer; Colorectal Neoplasms; Adenomatous Polyps; Adenoma; Advanced adenoma
MeSH Terms: conditions — Colorectal Neoplasms; Adenomatous Polyps; Adenoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case arm: Prospective enrollment of participants confirmed with colorectal adenocarcinoma or advanced adenoma
- Control arm: Prospective enrollment of healthy participants who have general risk or high risk of colorectal cancer

SUMMARY:
The primary objective of the study is to screen multi-omics markers in blood samples and construct a prediction model for CRC based on liquid biopsy, and we will further optimize the prediction model by validating its clinical performance externally.

DETAILED DESCRIPTION:
This multicenter research intends to enroll 3,600 participants according to predefined inclusion and exclusion criteria. The study will be divided into two groups: the "cancer arm" and the "control arm", with the "control arm" further subdivided into the "general-risk arm" and the "high-risk arm". All participants enrolled in this study will be required to provide a 10 ml whole blood sample.

This study consists of two sections. The first section involves constructing an diagnostic prediction model for early CRC detection, and the second section focuses on validating and optimizing this prediction model.

In the first section, a prediction model for the early detection of CRC will be developed with a cohort of 1,700 participants. This cohort comprises 900 individuals in the cancer arm, including 800 CRC patients and 100 with advanced adenoma (AA), along with 800 individuals in the control rm. All participants will be required to provide a 10 ml blood sample. Cell-free DNA (cfDNA) and microRNA (miRNA) will be sequenced and analyzed with the next-generation sequencing (NGS) platform,. And cancer specific markers will be identified to construct an early detection liquid biopsy prediction model by leveraging machine learning techniques and incorporating clinical pathological diagnostic information.

In the second section, a total of 1,900 participants were include, with 1,100 in the "cancer arm" (800 CRC and 300 AA patients) and 800 in the "control arm", the prediction model established in the first section will be validated in an external cohort, and algorithm optimization will be performed.

ELIGIBILITY:
Inclusion Criteria for Case Arm:

1. Aged over 18 years.
2. Participants confirmed with colorectal adenocarcinoma or advanced adenoma through colonoscopy and pathological examination.
3. Provision of informed consent prior to any study specific procedures, sampling, and analyses.

Inclusion Criteria for Control Arm:

1. Individuals of "General risk arm" should meet all the following criteria:

   1. No history of colorectal adenomas or sessile serrated polyps.
   2. No history of inflammatory bowel disease (8-10 years ).
   3. No family history (first-degree relatives) of colorectal cancer.
2. Individuals of "High-risk arm" should meet at least one of the following criteria:

   1. Asia-Pacific Colorectal Screening (APC) score ≥ 3.
   2. Family history (first-degree relatives) of colorectal cancer.
   3. History of positive fecal occult blood test.
   4. Any 2 of the following: chronic diarrhea, chronic constipation, mucous bloody stools, history of psychological stimulation, history of chronic appendicitis or appendectomy, history of chronic biliary disease or cholecystectomy.
   5. Individuals with inflammatory bowel disease.
3. All participants must be confirmed not to have colorectal malignancy or advanced adenomas through colonoscopy.
4. Provision of informed consent prior to any study specific procedures, sampling, and analyses.

Exclusion Criteria:

1. History of other malignant tumors (excluding non-melanoma skin cancer).
2. Prior or related treatments previously (including colorectal cancer or advanced adenoma surgery, endoscopic treatment, chemotherapy, targeted therapy, immunotherapy, radiation, neoadjuvant therapy, etc.).
3. Patients with hereditary colorectal diseases (including Lynch syndrome, familial CRC type X (FCCX), familial adenomatous polyposis (FAP), MUTHY-associated polyposis (MAP), Peutz-Jeghers syndrome (PJS), juvenile polyposis syndrome (JPS), serrated polyposis syndrome (SPS), etc.).
4. Usage of anti-tumor drugs such as methotrexate, cyclophosphamide, mercaptopurine, and bendamustine for other diseases within 30 days before blood collection.
5. Prior blood transfusion (including blood components) within the past 2 weeks.
6. Prior organ transplantation, bone marrow transplantation, or stem cell transplantation.
7. Pregnancy women.
8. Prior or current anti-infection treatment within 14 days before blood collection.
9. Inability to comply with study procedures such as blood collection and related examinations.
10. Deemed unsuitable for participation in the clinical trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Case arm: patients with colorectal cancer or advanced adenoma. Control arm: healthy participants who have general risk or high risk of colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 3600 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the screening test with comparison to colonoscopy | Through study completion, an average of 3 year
  Cancer specific markers will be identified to construct an early detection liquid biopsy prediction model, which will be compared with diagnostic colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Kefeng Ding, MD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (6):
- China (6):
  - The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Sun Yat-Sen University Cancer Hospital, Guangzhou
  - Yunnan cancer hospital, Kunming
  - Jiangsu province hospital, Nanjing
  - The first affiliated hospital of Xi'an Jiaotong University, Xi'an
  - Henan Cancer Hospital Affiliated Cancer Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No